CLINICAL TRIAL: NCT03343652
Title: A Phase I/II Clinical Trial to Evaluate the Safety and Efficacy of Nivolumab and Bendamustine Combination (NB) in Patients With Relapsed or Refractory Hodgkin's Lymphoma
Brief Title: A Study of Safety and Efficacy of Nivolumab and Bendamustine (NB) in Patients With Relapsed/Refractory Hodgkin's Lymphoma
Acronym: NB001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10/17-n
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Nivolumab; Bendamustine Hydrochloride
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NB (Experimental): Nivolumab 3 mg/kg IV infusion on day 1,14 + Bendamustine hydrochloride 90 mg/kg IV infusion on day 1,2 up to 3 cycles. Duration of cycle 28 days
  Interventions: Drug: Nivolumab; Drug: Bendamustine Hydrochloride

INTERVENTIONS:
Drug: Nivolumab — 3 mg/kg IV infusion on day 1,14 up to 3 cycles
  Other Names: Opdivo
Drug: Bendamustine Hydrochloride — 90 mg/kg IV infusion on day 1 up to 3 cycles
  Other Names: Ribomustin

SUMMARY:
A clinical study of safety and efficacy of treatment with Nivolumab and Bendamustine (NB) in patients with relapsed/refractory Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically confirmed Hodgkin's lymphoma
* Relapsed or refractory to at least two prior treatment lines
* Relapsed after nivolumab treatment or refractory to nivolumab treatment
* Age 18-70 years old
* Signed informed consent
* No severe concurrent illness

Exclusion Criteria:

* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent
* Active or prior documented autoimmune disease requiring systemic treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) of Nivolumab in combination with Bendamustine Hydrochloride in patients with Hodgkin's lymphoma | up to 3 months
  Overall response rate (ORR), defined as proportion of patients with complete response (CR) or partial response (PR) in measurable lesions as defined by LYRIC criteria and duration of response.

SECONDARY OUTCOMES:
Frequency of grade 3 or higher treatment-related adverse events by CTCAE 4.03 | up to 12 months
  Toxicity parameters based on NCI CTCAE 4.03 grades: hematological toxicity (CBC), hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), fatigue (attending physician assessment), rash (attending physician assessment), colitis (attending physician assessment), pneumonitis (attending physician assessment), autoimmune disorders (level of hormones, presence of autoimmune antibodies, attending physician assessment).
Duration of Response (DOR) | up to 12 months
  Duration of response will be measured from the time of initial response to nivolumab till documented disease progression, death or last evaluation of tumor status.
Time to Progression (TTP) | up to 12 months
Progression-Free Survival (PFS) | up to 12 months
Overall Survival (OS) | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Boris V Afanasyev, PhD, Study Director — First Pavlov State Medical University of St. Petersburg
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided